CLINICAL TRIAL: NCT05002829
Title: Complex And Simple Appendicitis: REstrictive or Liberal Post-operative Antibiotic eXposure (CASA RELAX) Using Desirability of Outcome Ranking (DOOR) and Response Adjusted for Duration of Antibiotic Risk (RADAR): A Randomized Controlled Trial at Denver Health
Brief Title: Restricted or Liberal Antibiotics After Appendectomy - Denver Health
Acronym: CASA RELAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Daniel Yeh, Professor of Surgery, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20191238
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Appendicitis
Keywords: post-operative; antibiotics
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restricted Post-Operative Antibiotics Group (Experimental): Participants undergoing standard of care (SOC) with simple appendicitis will not receive post-operative antibiotics.
  Participants undergoing standard of care with complicated (gangrenous or perforated) appendicitis will receive up to 24 hours of SOC post-operative antibiotics.
  Interventions: Other: Restricted Duration of SOC Antibiotic Use
- Liberal Post-Operative Antibiotics Group (Active Comparator): Participants undergoing standard of care with simple appendicitis will receive 24 hours of post-operative SOC antibiotics
  Participants undergoing standard of care with complicated (gangrenous or perforated) appendicitis will receive 4 days of post-operative SOC antibiotics.
  Interventions: Other: Liberal Duration of SOC Antibiotic Use

INTERVENTIONS:
Other: Restricted Duration of SOC Antibiotic Use — Standard of Care Antibiotic use will be restricted to none or up to 24 hours of post-operative antibiotics.
  Arms: Restricted Post-Operative Antibiotics Group
Other: Liberal Duration of SOC Antibiotic Use — Standard of Care Antibiotic use will be permitted for 24 hours or up to 4 days of post-operative antibiotics.
  Arms: Liberal Post-Operative Antibiotics Group

SUMMARY:
The purpose of this study is to see if decreasing the amount of antibiotics after appendicitis surgery can decrease the risk of adverse effects associated with antibiotics while at the same time ensuring participant safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Planned appendectomy (laparoscopic or open) for simple or complicated (perforated or gangrenous) appendicitis
* Working telephone number or reliable method to contact patient after hospital discharge

Exclusion Criteria:

* Unable to consent
* Pregnant Women
* Prisoners
* Immunocompromised as determined by clinical team, or patients actively receiving steroids, chemotherapy, or immunosuppressing medications (for example tacrolimus), or patients with active hematologic malignancy affecting the immune system, leukopenia, or end-stage AIDS
* Heart failure
* Allergy to bupivacaine
* Unlikely to comply with treatment or follow-up
* Inpatient consultation for appendicitis
* Clinically suspected of sepsis based on Sepsis-3 definition
* Current use of antibiotics for other indications
* Uncontrolled hyperglycemia or Type 1 Diabetes
* Surgeon preference
* Patient preference
* Research team unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with no antibiotic related adverse effects | Up to 40 days after appendicitis surgery
  As assessed by treating physician
Incidence of Infectious/Antibiotic Complications | Up to 30 days after appendicitis surgery
  Infectious/antibiotic complication requiring antibiotic treatment only, Emergency Department visit, hospital readmission, percutaneous drainage, and operative intervention as assessed by treating physician.
Number of participant deaths | Up to 30 days after appendicitis surgery
  As assessed by treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D Yeh, MD, MHPE, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sawyer RG, Claridge JA, Nathens AB, Rotstein OD, Duane TM, Evans HL, Cook CH, O'Neill PJ, Mazuski JE, Askari R, Wilson MA, Napolitano LM, Namias N, Miller PR, Dellinger EP, Watson CM, Coimbra R, Dent DL, Lowry SF, Cocanour CS, West MA, Banton KL, Cheadle WG, Lipsett PA, Guidry CA, Popovsky K; STOP-IT Trial Investigators. Trial of short-course antimicrobial therapy for intraabdominal infection. N Engl J Med. 2015 May 21;372(21):1996-2005. doi: 10.1056/NEJMoa1411162. PMID 25992746
- [Background] Yeh DD, Eid AI, Young KA, Wild J, Kaafarani HMA, Ray-Zack M, Kana'an T, Lawless R, Cralley AL, Crandall M; EAST Appendicitis Study Group. Multicenter Study of the Treatment of Appendicitis in America: Acute, Perforated, and Gangrenous (MUSTANG), an EAST Multicenter Study. Ann Surg. 2021 Mar 1;273(3):548-556. doi: 10.1097/SLA.0000000000003661. PMID 31663966
- [Background] Lawless RA, Cralley A, Qian S, Vasileiou G, Yeh DD; EAST Appendicitis Study Group. Antibiotics after Simple (Acute) Appendicitis are not Associated with Better Clinical Outcomes: A Post-Hoc Analysis of an EAST Multi-Center Study. Surg Infect (Larchmt). 2021 Jun;22(5):504-508. doi: 10.1089/sur.2019.348. Epub 2020 Sep 3. PMID 32897168
- [Background] Bou Zein Eddine S, Dodgion CM, Qian S, Trevino C, De Moya MA, Yeh DD; EAST Appendicitis Research Group. Complicated Appendicitis: Are Extended Antibiotics Necessary? A Post Hoc Analysis of the EAST Appendicitis "MUSTANG" Study. J Surg Res. 2020 Mar;247:508-513. doi: 10.1016/j.jss.2019.09.054. Epub 2019 Dec 4. PMID 31812337
- [Background] Evans SR, Rubin D, Follmann D, Pennello G, Huskins WC, Powers JH, Schoenfeld D, Chuang-Stein C, Cosgrove SE, Fowler VG Jr, Lautenbach E, Chambers HF. Desirability of Outcome Ranking (DOOR) and Response Adjusted for Duration of Antibiotic Risk (RADAR). Clin Infect Dis. 2015 Sep 1;61(5):800-6. doi: 10.1093/cid/civ495. Epub 2015 Jun 25. PMID 26113652
- [Derived] Yeh DD, Hatton GE, Pedroza C, Pust G, Mantero A, Namias N, Kao LS. Complex And Simple Appendicitis: REstrictive or Liberal postoperative Antibiotic eXposure (CASA RELAX) using Desirability of Outcome Ranking (DOOR) and Response Adjusted for Duration of Antibiotic Risk (RADAR): study protocol for a randomized controlled trial. Trauma Surg Acute Care Open. 2022 Sep 16;7(1):e000931. doi: 10.1136/tsaco-2022-000931. eCollection 2022. PMID 36148315